CLINICAL TRIAL: NCT06715189
Title: Correlation Between Serum Adiponectin and Resistin Levels and Degree of Hepatic Fibrosis In Metabolic Dysfunction _Associated Steatotic Liver Disease (MASLD)With Type2 Diabetes Mellitus
Brief Title: Correlation Between Serum Adiponectin And Resistin Levels And Degree of Hepatic Fibrosis in MASlD With type2 Diabetes Mellitus
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Elzahraa Kadry Mohamed, Teaching assistant fellow At sohag teaching hospital, Sohag University
Other Study IDs: Soh-Med-24-11--5MD
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Hepatic Fibrosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MASLD patients with hepatic fibrosis: MASLD with hepatic fibrosis with type 2 diabetes mellitus
  Interventions: Diagnostic Test: serum Adiponectine and Resistin; Diagnostic Test: fibroscan
- MASLD without hepatic fibrosis: MASLD with out hepatic fibrosis with type 2 diabetes mellutis
  Interventions: Diagnostic Test: serum Adiponectine and Resistin; Diagnostic Test: fibroscan

INTERVENTIONS:
Diagnostic Test: serum Adiponectine and Resistin — corrolation between serum adiponectin and Resistin levels and degree of hepatic fibrosis
Diagnostic Test: fibroscan — hepatic fibrosis detection in type 2 diabetes mellutis

SUMMARY:
Metabolic dysfunction asociated steatotic liver disease prevalence is 25%world wide diabetic patients have a risk for MASLD then have hepatic fibrosis so we study correlation Between Serum Adiponectin And Resistin Levels And Degree of Hepatic fibrosis In Metabolic dysfunction asociated steatotic liver disease in patients with type2 Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria:

* patients of both sex who have type2 Diabetes Mellitus for less than five years

Exclusion Criteria:alcholics ,chronic liver disease elevated liver functions , sever infection

-

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MASLD patients with hepatic fibrosis groupA,MASLD patients without hepatic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
degree of hepatic fibrosis in MASLD with type 2 diabetes mellitus | 1 year
  adiponectineand resistine level with degree of hepatic fibrosis in MASLD pt. with type 2 DM

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan WK, Chuah KH, Rajaram RB, Lim LL, Ratnasingam J, Vethakkan SR. Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD): A State-of-the-Art Review. J Obes Metab Syndr. 2023 Sep 30;32(3):197-213. doi: 10.7570/jomes23052. Epub 2023 Sep 13. PMID 37700494
- [Background] Marchesini G, Vettor R, Pinzani M. MASLD emerging from the fog of fatty liver. J Hepatol. 2024 Feb;80(2):178-180. doi: 10.1016/j.jhep.2023.10.011. Epub 2023 Nov 30. No abstract available. PMID 38278621
- [Background] Teng ML, Ng CH, Huang DQ, Chan KE, Tan DJ, Lim WH, Yang JD, Tan E, Muthiah MD. Global incidence and prevalence of nonalcoholic fatty liver disease. Clin Mol Hepatol. 2023 Feb;29(Suppl):S32-S42. doi: 10.3350/cmh.2022.0365. Epub 2022 Dec 14. PMID 36517002
- [Background] Estes C, Razavi H, Loomba R, Younossi Z, Sanyal AJ. Modeling the epidemic of nonalcoholic fatty liver disease demonstrates an exponential increase in burden of disease. Hepatology. 2018 Jan;67(1):123-133. doi: 10.1002/hep.29466. Epub 2017 Dec 1. PMID 28802062